CLINICAL TRIAL: NCT05979324
Title: Evaluation of the Effectiveness and Safety of ABAStroke in the Rehabilitation of Cognitive Deficits in Stroke Patients
Brief Title: Evaluation of the Effectiveness and Safety of ABAStroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ABAStroke Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABAStroke 1.0
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The intervention will take place over a maximum of 104 days, i.e. 15 weeks, a minimum of 13 weeks, i.e. 91 days. During this period, it is recommended to use the ABAstroke technology (app) for a maximum of 91 days along with standard therapy, including the possibility of using rehabilitation (as recommended by researchers or other physicians rehabilitating a patient after a stroke). The study is planned as a superiority study. Patients in the control group will be on standard stroke therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABAStroke Digital Therapeutics (Experimental): 50 patients using ABAStroke with standard treatment after a stroke.
  Interventions: Device: ABAStroke Digital Therapeutics
- Control group (No Intervention): 50 people using standard treatment after a stroke.

INTERVENTIONS:
Device: ABAStroke Digital Therapeutics — The total time of the study is 30 weeks in total, i.e. 15 weeks of patient recruitment and then a maximum of another 15 weeks until the end of the observation of the last patient. Within 2 weeks from the last patient, the last Monitor's visit will be performed to close the study. The patient will use the ABAStroke application for a maximum of 91 days (the minimum time is 28 days) and standard therapy, including rehabilitation (as recommended by researchers or other physicians rehabilitating a patient after a stroke).
  Arms: ABAStroke Digital Therapeutics

SUMMARY:
The aim of the project is to confirm the effectiveness and safety of the ABAStroke technology, which uses the principles of Applied Behavior Analysis (ABA) in the rehabilitation of cognitive deficits in patients after strokes. The study is comparative in nature, where a group of 100 patients will be included in this randomized study, divided equally into a study group and a control group. The purpose of the study is also to demonstrate that this non-invasive new rehabilitation technology based on the ABAStroke computer software supports the process of rehabilitation in the field of cognitive functions together with standard pharmacological therapy, including the possibility of using rehabilitation (as recommended by researchers and other doctors conducting rehabilitation of a patient after a stroke brain). ABAStroke can lead to improved cognitive functions (such as abstraction, short-term memory, visuospatial functions, executive functions, language, verbal fluency, allopsychic orientation, and attention) and is delivered via a mobile device app that can be used at home.

ELIGIBILITY:
Inclusion Criteria:

1. Men and/or women between the ages of 18 and 70
2. Condition after an ischemic or hemorrhagic stroke that occurred within the last 6 months before the start of the study.
3. MoCA score >14 and <26 points.
4. Signing of the informed consent form by each study participant.

Exclusion Criteria:

1. Vision disorders of various etiologies, which, in the opinion of the researcher, prevent the efficient use of a device using electronic displays.
2. Psychotic episodes and/or manic episodes and/or severe depression (Beck score 26 or higher) in the past year.
3. History of alcohol abuse or physical dependence on opioids in the past 2 years.
4. Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social circumstances) that could affect the patient's ability to attend scheduled appointments and use the investigational technology as determined by the investigator.
5. MoCA score <15 or >25 points.
6. Treatment of procognitive drug therapy in the last 6 months before inclusion in the study:

nootropics (pro-cognitive): cerebrolysin, citicoline, vinpocetine, nicergoline, piracetam, Gingo Biloba preparations, lecithin, cholinesterase inhibitors: donepezil, rivastigmine, galantamine, NMDA receptor antagonist: memantine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
MoCA | 3 months
  Screening tool for detecting cognitive deficits

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Neurology of the Jagiellonian University Hospital, Krakow, Poland